CLINICAL TRIAL: NCT07185061
Title: Clinical Study on Acoustic Stimulation Intervention in Chronic Tinnitus Patients
Brief Title: Interventional Treatment of Chronic Tinnitus With Acoustic Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-SR-547
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2024-10

CONDITIONS: Chronic Tinnitus
MeSH Terms: interventions — Acoustic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic tinnitus (Experimental)
  Interventions: Device: Acoustic Stimulation

INTERVENTIONS:
Device: Acoustic Stimulation — Using hearing loss detection and tinnitus matching data as input parameters, the system automatically generates personalized sound stimulation audio signals through composite signal amplitude, frequency, phase control processing, and notch filtering. The audio tone is fine-tuned based on the patient's initial treatment response to identify their most comfortable range.

SUMMARY:
The《Clinical practice guideline: tinnitus》defines tinnitus as the perception of sound without an external source, with patients lasting six months or longer classified as chronic tinnitus. Epidemiological studies indicate that tinnitus affects up to 25% of the global population. With a worldwide estimated 7.2 billion people affected, which translates to approximately 1.8 billion individuals impacted. Among these, 33% (about 590 million people) experience varying degrees of hearing impairment, and severely disrupting their work, daily life, and social interactions. Furthermore, 10%-15% of patients (approximately 180～270 million) require medical treatment or intervention. Notably, tinnitus prevalence increases with age: it affects about 29.7% of those over 60 and rises to 33% for those aged 65 and above. These statistics demonstrate that tinnitus has become one of the most significant global health challenges.

In recent years, many studies have proposed an innovative therapeutic approach for tinnitus based on new research advancements in its pathogenesis. The methods termed Active Tinnitus Stimulation Therapy (ATST) and focuses on central mechanisms of tinnitus, abnormal neuronal discharges, and neural plasticity in related brain regions. The therapy tailors acoustic stimulation protocols according to individual hearing loss severity and tinnitus characteristics. Specifically, tailored acoustic signals are converted into electrical impulses in the cochlea, transmitted through auditory pathways to thalamic and auditory cortex nuclei. This process actively modulates auditory pathways, enhances filtering of chaotic signals, and activates auditory neurons. By synchronizing the self-discharge of neurons with nearby captured sound signals, ATST disrupts tinnitus generation and suppresses amplification, thereby reducing patients 'perception of tinnitus sounds. The approach comprehensively analyzes patients' hearing thresholds and tinnitus characteristics to generate personalized acoustic stimuli. Through targeted neuronal stimulation, it regulates neural plasticity, reduces abnormal discharges, and achieves active neuromodulation. Although some studies suggest that long-term periodic acoustic stimulation therapy may weaken tinnitus-related EEG networks, indicating potential improvement in chronic tinnitus, there remains a lack of large-scale clinical evidence confirming the effectiveness of this treatment for chronic tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic tinnitus lasting over six months (with or without hearing loss), showing no organic lesions in the auditory conduction pathway or temporal bone, and either not receiving any treatment (including medication or traditional Chinese medicine) or having discontinued therapy for over three months. These patients must be mentally alert, mentally stable, and able to provide fluent responses to all questions from the doctor and research team members.

Exclusion Criteria:

* Patients with organic lesions in the auditory conduction pathway and temporal bone (e.g., tympanic membrane perforation, ossicular chain disruption), other otological conditions such as Meniere's disease, vertigo, chronic otitis media, middle ear cholesteatoma, or acute/chronic external otitis, history of head trauma or central nervous system disorders, exposure to ototoxic drugs, use of tinnitus medications or traditional Chinese medicine treatments (within 3 months of discontinuation), inability to cooperate with medical procedures or answer questions, or participants who dropped out or lost contact within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Scores of Tinnitus Handicap Inventory | From enrollment to the end of treatment at 12 weeks

SECONDARY OUTCOMES:
Scores of Self-rating Anxiety Scale | From enrollment to the end of treatment at 12 weeks
Scores of Pittsburgh sleep quality index | From enrollment to the end of treatment at 12 weeks
Scores of Self-ratingDepression Scale | From enrollment to the end of treatment at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No